CLINICAL TRIAL: NCT00740909
Title: Cognitive Behavioral Therapy for Trichotillomania
Acronym: CBT for TTM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Nancy J. Keuthen, Nancy J. Keuthen, Ph.D, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008P000565
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Trichotillomania
Keywords: Trich; Hair Pulling; Cognitive Behavioral Therapy; Behavioral Therapy
MeSH Terms: conditions — Trichotillomania; Trichomonas Infections | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- MAC (No Intervention): Minimal Attention Control
- CBT (Experimental): Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — A therapy designed to help patients with response prevention skills.
  Arms: CBT

SUMMARY:
This study aims to develop a comprehensive Cognitive Behavioral Therapy protocol for adult patients with Trichotillomania that emphasizes relapse prevention and that addresses comorbid affective symptoms, as well. The study will compare the efficacy of CBT with a minimal attention control (MAC)condition. We hypothesize that outcome at post-treatment, 3-month, and 6-month follow-up will be better for the CBT vs. MAC condition including higher responder rates and greater reduction in hair pulling severity.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of cognitive behavioral therapy for patients with trichotillomania.

Following entry into the study, subjects will be randomized into a cognitive behavioral therapy (CBT) or a minimized attention control (MAC) condition. Subjects will be assessed with the Acceptance and Action Questionnaire (AAQ), the Affective Regulation Rating (ARR), the Barratt Impulsivity Scale (BIS-11), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), Clinical Global Impressions Scale (CGI), the Difficulties in Emotion Regulation Scale (DERS), Hair Pulling Scale (HPS), Trichotillomania (TTM) Impact Scale, Psychiatric Institute Trichotillomania Scale (PITS), National Institute of Mental Health Trichotillomania Severity Scale(NIMH-TSS), the Generalized Expectancy for Negative Mood Regulation Scale (NMR), The Milwaukee Inventory for Subtypes of Trichotillomania- Adult Version (MIST-A), the Positive and Negative Affect Scale (PANAS), the Quality of Life Inventory (QOLI), the Readiness to Change Hairpulling Behavior (RCHPB), the Self-Esteem Scale (SES), the Skin Picking Scale (SPS) and the Scales of Psychological Well-Being (SPWB). Subject randomization to a treatment arm will be determined by a random number generator.

Subject change scores will be assessed for the above scales.

ELIGIBILITY:
Inclusion Criteria:

* primary DSM-IV diagnosis of TTM
* outpatients who are 18 or older
* a minimum MGHHPS total scale score of 10
* a minimum TTM symptom duration of 1 year with no significant remissions (as defined by complete abstinence of hair extraction for a 2-week period during the prior 6 months)

Exclusion Criteria:

* presence of a serious psychiatric condition including mental retardation, psychosis, pervasive developmental disorder, organic mental disorders, manic episode, ADHD, suicidality, lifetime alcohol or substance dependence, or alcohol or substance abuse within the past 3 months
* presence of a serious medical condition that would limit ability to routinely attend sessions and complete homework assignments
* individual or group psychotherapy (not addressing TTM) that has not been ongoing for the past 3 months and/or without intent to continue same treatment during study tenure)
* previous CBT for TTM
* involvement in other treatment for TTM
* psychotropic medication that has not been stable for 3 months prior to study enrollment and/or without intent to continue same medication regimen during study tenure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Massachusetts General Hospital Hair Pulling Scale (MGHHPS) | Baseline, weekly visits, follow-up
NIMH Trichotillomania Severity Scale (NIMH-TSS) | Baseline, weekly visits, follow-up
NIMH Trichotillomania Impairment Scale (NIMH-TIS) | Baseline, weekly visits, follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Keuthen, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Keuthen NJ, Rothbaum BO, Falkenstein MJ, Meunier S, Timpano KR, Jenike MA, Welch SS. DBT-enhanced habit reversal treatment for trichotillomania: 3-and 6-month follow-up results. Depress Anxiety. 2011 Apr;28(4):310-3. doi: 10.1002/da.20778. Epub 2010 Dec 15. PMID 21456040